CLINICAL TRIAL: NCT01303068
Title: Detection of Pseudomonas. Aeruginosa in the Airways of Patients With Cystic Fibrosis Using of Aerosolized 13C-urea
Brief Title: Detection of Pseudomonas Aeruginosa in the Airways of Patients With CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Hengameh Raissy, Pharm.D., Research Associate Professor, Pediatrics, University of New Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HRRC, 12-521
Record Dates: First submitted 2011-02-14; First posted 2011-02-24 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CF patients, 13C urea breath test kit (Experimental): CF patients with Pseudomonas infection tested with 13C urea breath test
  Interventions: Device: 13C urea breath test Kit
- Healthy controls, 13C urea breath test kit (Active Comparator): Healthy subjects using 13C urea breath test kit
  Interventions: Device: 13C urea breath test Kit

INTERVENTIONS:
Device: 13C urea breath test Kit — 20 and 50 mg, 13C urea breath test: urea nebulizer solution to detect Pseudomonas

SUMMARY:
The purpose of this study is to determine if inhaled urea can be used to detect the presence of Pseudomonas Aeruginosa in the lungs

DETAILED DESCRIPTION:
Dose Escalation study

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF aged 18 years and above colonized with P. aeruginosa
* Normal subjects ages 18 and above without CF or p. aeruginosa

Exclusion Criteria:

* for patients and volunteers will include the presence of asthma, allergic rhinitis, pregnancy, a history of gastric or duodenal ulcer, smoking, and a baseline FEV1 less than 60% of predicted normal value and a pulmonary exacerbation within the last 2 weeks as defined by use of systemic antibiotic

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08-15 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hengameh Raissy, PharmD, Principal Investigator — UNM
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subjects Using 13C Urea Breath Test Kit: Healthy subjects using 13C urea breath test kit
  13C urea breath test Kit: 20 and 50 mg, 13C urea breath test: urea nebulizer solution to detect Pseudomonas
Period: Overall Study
Arm/Group | CF Patients, 13C Urea Breath Test Kit | Healthy Subjects Using 13C Urea Breath Test Kit
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF Patients, 13C Urea Breath Test Kit | Healthy Controls, 13C Urea Breath Test Kit | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 26 [23 to 31] | 32 [24 to 41] | 29 [23 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective is to Assess the Safety of 13C Urea Administered by Inhalation.
Description: The primary endpoint is the safety of inhaled 13C urea assessed by adverse events including pulmonary findings and changes from baseline in physical examination findings, pulse oximetry results, pulmonary function test results, and vital signs.
Time Frame: 6 hours
Measure: Number; unit: adverse events
Arm/Group | CF Patients, 13C Urea Breath Test Kit | Healthy Subjects Using 13C Urea Breath Test Kit
Number analyzed (Participants) | 6 | 6
adverse events | 0 | 0

2. Secondary Outcome: The Secondary Objective is to Assess the Kinetics of 13C Carbon Dioxide Production by Measuring the Isotopic Ratio of 13C to 12C in Exhaled Carbon Dioxide.
Description: Secondary endpoints are the isotopic ratios of 13C to 12C in exhaled carbon dioxide measured with the POCone detector (Meretek Diagnostics Group of Otsuka America Pharmaceutical, Rockville, MD) at 5, 10, and 15 minutes after study drug administration.
Time Frame: 5 minutes post inhalation
Population: CF patients with infection has a higher 13C urea in their exhaled breath.
Measure: Mean (Full Range); unit: ratio
Arm/Group | CF Patients, 13C Urea Breath Test Kit | Healthy Subjects Using 13C Urea Breath Test Kit
Number analyzed (Participants) | 6 | 6
ratio
  20 mg: number analyzed (Participants) | 3 | 3
  20 mg | 4 [2.2 to 4.9] | 0.8 [0.4 to 1.2]
  50 mg: number analyzed (Participants) | 3 | 3
  50 mg | 10 [6.2 to 14.5] | 2.13 [0.1 to 5.5]

ADVERSE EVENTS:
Arm/Group | CF Patients, 13C Urea Breath Test Kit | Healthy Subjects Using 13C Urea Breath Test Kit
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-11-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT01303068/Prot_000.pdf
  • Informed Consent Form (2012-11-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT01303068/ICF_001.pdf